CLINICAL TRIAL: NCT01974999
Title: A Retrospective Multicenter Study to Determine 5-Year Clinical Outcomes in Subjects Previously Enrolled in the CTOT-01 Study (CTOT-17)
Brief Title: A Retrospective Multicenter Study to Determine 5-Year Clinical Outcomes in Subjects Previously Enrolled in the CTOT-01 Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-17
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Kidney Disease; Kidney Failure; End Stage Renal Disease
Keywords: Kidney; Transplant; Rejection
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Kidney Failure, Chronic; Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a multicenter, non-randomized, retrospective study to collect long term (5 years post-transplant) clinical outcome data to test whether the results of the noninvasive immune monitoring test strategy performed in the parent study (CTOT-01, NCT00308802) in first six-month post-transplant is predictive of 5-year outcomes. Each center will complete a retrospective chart review for the data on patient survival, graft survival and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Participants previously enrolled in the CTOT-01 study.
* Participants who are at least 5 years post-transplant (+/- 6 months), no later than March 31, 2014.

Exclusion Criteria:

* Withdrawal of consent to continue in the CTOT-01 study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was selected based on their previous participation in the parent study (CTOT-01). A total of 280 subjects were enrolled and transplanted in the Clinical Trials in Organ Transplantation
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration Rate (eGFR) from 6 months to 5 years post-transplantation | Day 1
  Modification of Diet in Renal Disease (MDRD) in the adult cohort and Schwartz method in the pediatric cohort

SECONDARY OUTCOMES:
Patient survival as assessed by the incidence of death reported in the first 5 years post- transplant | Day 1
Graft survival as assessed by the incidence of graft loss reported in the first 5 years post- transplant | Day 1
Renal function as assessed by the absolute glomerular filtration Rate (GFR) at 5 years post-transplant | Day 1
Change in Chronic Kidney Disease stages between transplant and 5 years post- transplant | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Donald E Hricik, MD, Study Chair — University Hospitals Cleveland Medical Center
Locations (7):
- United States (5):
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Glickman Urological Institute, Cleveland, Ohio
- Canada (2):
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba

REFERENCES:
- [Result] Faddoul G, Nadkarni GN, Bridges ND, Goebel J, Hricik DE, Formica R, Menon MC, Morrison Y, Murphy B, Newell K, Nickerson P, Poggio ED, Rush D, Heeger PS; CTOT-17 consortium. Analysis of Biomarkers Within the Initial 2 Years Posttransplant and 5-Year Kidney Transplant Outcomes: Results From Clinical Trials in Organ Transplantation-17. Transplantation. 2018 Apr;102(4):673-680. doi: 10.1097/TP.0000000000002026. PMID 29189482
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) — http://www.ctotstudies.org/
- Available data/document: Individual Participant Data Set: SDY1094 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY1094 — Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. Data analysis tools are also available to researchers.
- Available data/document: Study Protocol: SDY1094 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY1094 — ImmPort study identifier is SDY1094.
- Available data/document: Study summary, -design, -summary of participant assessments, -interventions, -medications, -demographics, -lab tests, -study files et al.: SDY1094 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY1094 — ImmPort study identifier is SDY1094.